CLINICAL TRIAL: NCT01062568
Title: The Adrenal Contribution to Androgen Production in Girls During Puberty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jeffrey Chang, MD, Principal Investigator, University of California, San Diego
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 091676
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Development
Keywords: adolescents; puberty; androgens; hyperandrogenemia
MeSH Terms: interventions — Adrenocorticotropic Hormone; Cosyntropin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obese group (Experimental): Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take a single oral dose of dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood sample drawn for hormone measurements. After this blood sample, adrenocorticotropin (ACTH) will be administered as an iv bolus. At 30 and 60 minutes after ACTH, blood samples will be obtained for repeat hormone measurements.
  Interventions: Drug: Adrenocorticotropin; Drug: Dexamethasone
- Nonobese group (Experimental): Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take a single oral dose of dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood sample drawn for hormone measurements. After this blood sample, adrenocorticotropin (ACTH) will be administered as an iv bolus. At 30 and 60 minutes after ACTH, blood samples will be obtained for repeat hormone measurements.
  Interventions: Drug: Adrenocorticotropin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Adrenocorticotropin — Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take a single oral dose of dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood sample drawn for hormone measurements. After this blood sample, adrenocorticotropin (ACTH) will be administered as an iv bolus. At 30 and 60 minutes after Cosyntropin, blood samples will be obtained for repeat hormone measurements.
  Other Names: Cosyntropin; ACTH
Drug: Dexamethasone — Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take a single oral dose of dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood sample drawn for hormone measurements. After this blood sample, 0.25 mg adrenocorticotropin (ACTH) will be administered as an iv bolus. At 30 and 60 minutes after Cosyntropin, blood samples will be obtained for repeat hormone measurements.
  Other Names: dex

SUMMARY:
In girls with elevated androgens the precise source of androgen excess throughout puberty and early adolescence has not been carefully examined. The investigators propose to examine whether the adrenal gland produces the majority of androgens during puberty by studying the differences in androgen responses to adrenocorticotropin hormone (ACTH) administration in normal weight (NW) and obese (OB) girls ages 7-18. The investigators' analyses will compare steroid changes before and 60 min after ACTH administration in NW and OB girls.

DETAILED DESCRIPTION:
Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take a single oral dose of dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood sample drawn for hormone measurements. After this blood sample, 0.25 mg adrenocorticotropin hormone (ACTH) will be administered as an iv bolus. At 30 and 60 minutes after Cosyntropin, blood samples will be obtained for repeat hormone measurements.

ELIGIBILITY:
Inclusion Criteria:

* Normal CBC (Hemoglobin must be at least 11mg/dl)
* Normal renal and liver function tests (AST& ALT 10-45 IU/L; Albumin 3.3-5 g/dL; Alk phos 30-130 IU/L;
* direct bili <0.2 mg/dL;
* total bili <1.2 mg/dL; total protein 6.0-8.0 g/dL) Normal vital signs including normal blood pressure (pulse 60-100/min, respirations 12-20/min, BP 80/60-130/80)

Exclusion Criteria:

* Pregnancy
* On oral contraceptives
* On insulin lowering drugs
* On anti-androgens (i.e., spironolactone, flutamide, finasteride, etc)
* On medications that will influence androgen metabolism or clearance
* On medications that will inhibit the cytochrome P450 enzyme system (cimetidine, ketoconazole, etc)
* Subjects with morning cortisol<5 ug/dL will be excluded and asked to see their primary care physician.
* Subjects with 17-OHP>250 ng/dL) will be excluded and asked to see their primary care physician.
* Subject with a history of Cushing syndrome or adrenal insufficiency will be excluded

Ages: 7 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R J Chang, MD, Principal Investigator — UCSD
Locations (1):
- University of california, san diego, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Puberty Group: Subjects were subdivided into normal weight and overweight groups. Blood was drawn at 1900 hr for baseline measurements. At 2200 hr each subject will take dexamethasone. At 0700 hr the following day, subjects will have a blood drawn for hormone measurements. After this adrenocorticotropin (ACTH) will be administered. At 30 and 60 minutes after ACTH, blood will be obtained for repeat hormone measurements.
  Adrenocorticotropin: Subjects will have blood drawn at 1900 hr for baseline measurements. At 2200 hr each subject will take a oral dose of dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood drawn for hormone measurements. After this blood sample, adrenocorticotropin (ACTH) will be administered. At 30 and 60 minutes after Cosyntropin, blood will be obtained for repeat hormone measurements.
- Late Puberty Group: Subjects were subdivided into normal weight and overweight groups. Subjects will have blood drawn at 1900 hr for baseline measurements. At 2200 hr each subject will take dexamethasone. At 0700 hr the following day, subjects will have a blood drawn for hormone measurements. After this adrenocorticotropin (ACTH) will be administered. At 30 and 60 minutes after ACTH, blood will be obtained for repeat hormone measurements.
  Adrenocorticotropin: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take dexamethasone. At 0700 hr the following day, subjects will have a blood drawn for hormone measurements. After this blood sample, adrenocorticotropin (ACTH) will be administered. At 30 and 60 minutes after Cosyntropin, blood samples will be obtained for repeat hormone measurements.
  Dex
Period: Overall Study
Arm/Group | Early Puberty Group | Late Puberty Group
Started | 10 | 40
Completed | 10 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Early Puberty Group: Subjects were subdivided into normal weight and overweight groups. Subjects will have blood drawn at 1900 hr for baseline measurements. At 2200 hr each subject will take dexamethasone. At 0700 hr the following day, subjects will have a blood drawn for hormone measurements. After this adrenocorticotropin (ACTH) will be administered as an iv bolus. At 30 and 60 minutes after ACTH, blood will be obtained for repeat hormone measurements.
  Adrenocorticotropin: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take a oral dose of dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood drawn for hormone measurements. After this, adrenocorticotropin (ACTH) will be administered. At 30 and 60 minutes after Cosyntropin, blood samples will be obtained for repeat hormone measurements.
  Dex
- Late Puberty Group: Subjects were further subdivided into normal weight and overweight groups. Subjects will have blood drawn at 1900 hr for baseline measurements. At 2200 hr each subject will take dexamethasone. At 0700 hr the following day, subjects will have a blood drawn for hormone measurements. After this, adrenocorticotropin (ACTH) will be administered. At 30 and 60 minutes after ACTH, blood will be obtained for repeat hormone measurements.
  Adrenocorticotropin: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood drawn for hormone measurements. After this, adrenocorticotropin (ACTH) will be administered as an iv bolus. At 30 and 60 minutes after Cosyntropin, blood samples will be obtained for repeat hormone measurements.
  Dex
- Total: Total of all reporting groups
Arm/Group | Early Puberty Group | Late Puberty Group | Total
Number analyzed (Participants) | 10 | 40 | 50
Age, Continuous [Mean (Standard Deviation); unit: years]
  Normal Wieght | 9.8 (1) | 13.9 (0.9) | 12.1 (1)
  Overweight | 9.4 (0.7) | 14.9 (0.4) | 12.4 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 40 | 50
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: 17-hydroxyprogesterone Response to ACTH
Description: 17-hyrooxyprogesterone levels before and after ACTH
Time Frame: 0 and 60 minutes after ACTH administration
Population: Analysis is performed on a normal weight group comprised of 4 early puberty and 10 late puberty girls and an overweight group of 6 early puberty and 30 late puberty girls
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Early Puberty Group; Late Puberty Group: Subjects were further subdivided into normal weight and overweight groups. Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take a single oral dose of dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood sample drawn for hormone measurements. After this blood sample, adrenocorticotropin (ACTH) will be administered as an iv bolus. At 30 and 60 minutes after ACTH, blood samples will be obtained for repeat hormone measurements.
- Total Number: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take a single oral dose of dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood sample drawn for hormone measurements. After this blood sample, adrenocorticotropin (ACTH) will be administered as an iv bolus. At 30 and 60 minutes after ACTH, blood samples will be obtained for repeat hormone measurements.
  Adrenocorticotropin: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take a single oral dose of dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood sample drawn for hormone measurements. After this blood sample, adrenocorticotropin (ACTH) will be administered as an iv bolus. At 30 and 60 minutes after Cosyntropin, blood samples will be obtained for repeat hormone measurements.
  Dex
Arm/Group | Early Puberty Group | Late Puberty Group | Total Number
Number analyzed (Participants) | 10 | 40 | 50
ng/mL
  Normal Weight: number analyzed (Participants) | 4 | 10 | 14
  Normal Weight | 2.4 (0.5) | 3.7 (0.8) | 3.1 (0.6)
  Over Weight: number analyzed (Participants) | 6 | 30 | 36
  Over Weight | 2.9 (0.4) | 3.1 (0.7) | 3.0 (0.6)

2. Secondary Outcome: Free Testosterone Response to ACTH
Description: Free Testosteorne levels before and after ACTH
Time Frame: 0 and 60 min after ACTH administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pmol/L
Groups:
- Early Puberty Group; Late Puberty Group: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take dexamethasone. At 0700 hr the following day, subjects will have a blood drawn for hormone measurements. After this, adrenocorticotropin (ACTH) will be administered. At 30 and 60 minutes after ACTH, blood will be obtained for repeat hormone measurements.
  Adrenocorticotropin: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take dexamethasone. At 0700 hr the following day, subjects will have a blood drawn for hormone measurements. After this , adrenocorticotropin (ACTH) will be administered. At 30 and 60 minutes after Cosyntropin, blood will be obtained for repeat hormone measurements.
Arm/Group | Early Puberty Group | Late Puberty Group
Number analyzed (Participants) | 10 | 40
pmol/L
  Normal weight: number analyzed (Participants) | 4 | 10
  Normal weight | 2 (0.3) | 7 (1)
  Overweight: number analyzed (Participants) | 6 | 30
  Overweight | 3.5 (0.4) | 32 (3)

3. Secondary Outcome: Androstenedione Response to ACTH
Description: Androstenedione levels before and after ACTH
Time Frame: 0 and 60 min after ACTH administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Early Puberty: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take dexamethasone. At 0700 hr the following day, subjects will have a blood drawn for hormone measurements. After this, adrenocorticotropin (ACTH) will be administered. At 30 and 60 minutes after ACTH, blood will be obtained for repeat hormone measurements.
  Adrenocorticotropin: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take dexamethasone. At 0700 hr the following day, subjects will have a blood drawn for hormone measurements. After this , adrenocorticotropin (ACTH) will be administered. At 30 and 60 minutes after Cosyntropin, blood will be obtained for repeat hormone measurements.
- Late Puberty: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take dexamethasone. At 0700 hr the following day, subjects will have a blood drawn for hormone measurements. After this , adrenocorticotropin (ACTH) will be administered. At 30 and 60 minutes after ACTH, blood will be obtained for repeat hormone measurements.
  Adrenocorticotropin: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take dexamethasone . At 0700 hr the following day, subjects will have a blood drawn for hormone measurements. After this, adrenocorticotropin (ACTH) will be administered. At 30 and 60 minutes after Cosyntropin, blood samples will be obtained for repeat hormone measurements.
Arm/Group | Early Puberty | Late Puberty
Number analyzed (Participants) | 10 | 40
ng/mL
  Normal Wieght: number analyzed (Participants) | 4 | 10
  Normal Wieght | 0.5 (0.1) | 1.6 (0.3)
  Overweight: number analyzed (Participants) | 6 | 30
  Overweight | 0.6 (0.2) | 3.1 (0.7)

ADVERSE EVENTS:
Groups:
- Early Puberty: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take a single oral dose of dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood sample drawn for hormone measurements. After this blood sample, adrenocorticotropin (ACTH) will be administered as an iv bolus. At 30 and 60 minutes after ACTH, blood samples will be obtained for repeat hormone measurements.
  Adrenocorticotropin: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take a single oral dose of dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood sample drawn for hormone measurements. After this blood sample, adrenocorticotropin (ACTH) will be administered as an iv bolus. At 30 and 60 minutes after Cosyntropin, blood samples will be obtained for repeat hormone measurements.
  .
- Late Puberty: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take a single oral dose of dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood sample drawn for hormone measurements. After this blood sample, adrenocorticotropin (ACTH) will be administered as an iv bolus. At 30 and 60 minutes after ACTH, blood samples will be obtained for repeat hormone measurements.
  Adrenocorticotropin: Subjects will have blood drawn at 1900 hr for baseline hormone measurements. At 2200 hr each subject will take a single oral dose of dexamethasone at 2200 hr. At 0700 hr the following day, subjects will have a blood sample drawn for hormone measurements. After this blood sample, adrenocorticotropin (ACTH) will be administered as an iv bolus. At 30 and 60 minutes after Cosyntropin, blood samples will be obtained for repeat hormone measurements.
Arm/Group | Early Puberty | Late Puberty
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/40
Other Adverse Events (participants affected / at risk) | 0/10 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No